CLINICAL TRIAL: NCT01254370
Title: A Phase 2, Randomized Study Evaluating the Safety and Efficacy of Catioprost® (Unpreserved Latanoprost 0.005% Emulsion) Compared to Travatan Z® in Subjects With Glaucoma or Ocular Hypertension and Ocular Surface Disease
Brief Title: Safety and Efficacy Study of Catioprost® (Unpreserved Latanoprost 0.005% Emulsion) Compared to Travatan Z® to Treat Glaucoma and Ocular Surface Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NVG10E118
Record Dates: First submitted 2010-11-29; First posted 2010-12-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: Glaucoma; Ocular Hypertension; Ocular Surface Disease
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost; Travoprost

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Catioprost (Experimental)
  Interventions: Drug: Latanoprost
- Travatan Z (Active Comparator)
  Interventions: Drug: Travatan Z

INTERVENTIONS:
Drug: Latanoprost — 0.005%
  Arms: Catioprost
Drug: Travatan Z — 0.004%
  Arms: Travatan Z

SUMMARY:
The purpose of this study is to compare:

* the effect of Catioprost® and Travatan Z® on the ocular surface disease (OSD) in subjects with glaucoma or ocular hypertension and ocular surface disease.
* the intraocular pressure (IOP) lowering effect and safety of Catioprost® and Travatan Z® in subjects with glaucoma or ocular hypertension and ocular surface disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age at Visit 1 (IOP Screening), of either sex and any race or ethnicity.
* Be willing and able to provide written informed consent prior to any study procedures being performed.
* Be willing and able to follow all instructions and attend all study visits.
* Have a documented diagnosis of ocular hypertension, open angle glaucoma (with or without pseudoexfoliation or pigment dispersion component) or chronic angle closure glaucoma with a patent iridotomy requiring treatment with an ocular hypertensive therapy in the study eye.
* Agree to submit to a pregnancy test at Visit 1 and at Visit 4, or not be of childbearing potential.
* Agree to use an acceptable method of contraception for the duration of the study or not be of childbearing potential. Acceptable methods of birth control include: spermicide with barrier, oral, transdermal, injectable, or implantable contraception, IUD, abstinence, and surgical sterilization of partner. Female subjects are not of childbearing potential if they have had a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or are post-menopausal by at least 12 months.

Exclusion Criteria:

* Have known sensitivity or poor tolerance to latanoprost or travoprost or any other component of the study medications.
* Have any form of glaucoma other than open angle glaucoma (with or without a pigment dispersion or pseudoexfoliation component), ocular hypertension or chronic angle closure glaucoma with patent iridotomy in either eye.
* Have an IOP at any time point during the Screening or Baseline visits (Visits 1 or 2) of > 34 mmHg in either eye.
* Be currently pregnant, nursing, or planning a pregnancy during the study period; or be a woman that has a positive pregnancy test.
* Have a history of any significant ocular condition(s) in either eye that would contraindicate the use of latanoprost or travoprost, or that might affect the study conduct or the interpretation of the study results.
* Have any abnormality preventing reliable Goldmann applanation tonometry of either eye.
* Have been previously non-responsive to prostaglandin analog therapy for reduction of IOP.
* Have prior (within 30 days of Visit 1) or anticipated concurrent use of an investigational drug or device during the study period.
* Have a condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of Catioprost versus Travatan Z | 3 months
  Efficacy measures:
  * Change from baseline in Intraocular Pressure (IOP)
  * Change in Ocular Surface Disease (OSD)

CONTACTS AND LOCATIONS:
Locations (1):
- Ora (Ophthalmic Research Associates), Andover, Massachusetts, United States